CLINICAL TRIAL: NCT02175017
Title: ONO-4538 Multicenter, Open-label, Uncontrolled, Phase II Study in Advanced Non-small Cell Lung Cancer
Brief Title: ONO-4538 Study in Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4538-09
Record Dates: First submitted 2014-06-18; First posted 2014-06-26 (Estimated); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-04

CONDITIONS: Advanced Non-small Cell Lung Cancer (NSCLC)
Keywords: ONO-4538; Advanced non-small cell lung cancer (NSCLC); nivolumab
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ONO-4538 for squamous non-small-cell lung cancer (NSCLC) (Experimental): In each treatment cycle, patients received an intravenous infusion of nivolumab (ONO-4538) at a dose of 3 mg/kg every 2 weeks for 6 weeks. Changes in dose were not allowed. Radiological assessments (computed tomography/ magnetic resonance imaging) were conducted every 6 weeks. Patients entered subsequent treatment cycles unless they met discontinuation criteria, including disease progression, unacceptable adverse events, and consent withdrawal. Patients who were discontinued for any of these reasons entered the follow-up phase.
  Interventions: Drug: ONO-4538
- ONO-4538 for non-squamous non-small-cell lung cancer (NSCLC) (Experimental): In each treatment cycle, patients received an intravenous infusion of nivolumab (ONO-4538) at a dose of 3 mg/kg every 2 weeks for 6 weeks. Changes in dose were not allowed. Radiological assessments (computed tomography/ magnetic resonance imaging) were conducted every 6 weeks. Patients entered subsequent treatment cycles unless they met discontinuation criteria, including disease progression, unacceptable adverse events, and consent withdrawal. Patients who were discontinued for any of these reasons entered the follow-up phase.
  Interventions: Drug: ONO-4538

INTERVENTIONS:
Drug: ONO-4538 — ONO-4538 Study in Patients With Squamous NSCLC
  Other Names: nivolumab
  Arms: ONO-4538 for squamous non-small-cell lung cancer (NSCLC)
Drug: ONO-4538 — ONO-4538 Study in Patients With Non-Squamous NSCLC
  Other Names: nivolumab
  Arms: ONO-4538 for non-squamous non-small-cell lung cancer (NSCLC)

SUMMARY:
The objective of the study is to investigate the efficacy and safety of ONO-4538 in subjects with stage IIIB/IV or recurrent non-small cell lung cancer unsuited to radical radiotherapy and resistant to a platinum-based chemotherapeutic regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 20 years of age
2. Histologically or cytologically confirmed non-small cell lung cancer
3. Diagnosis of NSCLC in stage IIIB/IV unsuited to radical radiotherapy according to UICC-TNM classification (7th edition) or recurrent NSCLC
4. Has at least one measurable lesion, as defined by the RECIST guideline (version 1.1)

Exclusion Criteria:

1. Current or prior severe hypersensitivity to another antibody product
2. Multiple primary cancers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2021-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitsunobu Tanimoto, Study Director — Ono Pharmaceutical Co. Ltd
Locations (10):
- South Korea (10):
  - Goyang-si Clinical Site 103, Goyang-si, Gyeonggi-do
  - Seongnam-si Clinical Site 104, Seongnam-si, Gyeonggi-do
  - Cheongju-si Clinical Site 106, Cheongju-si, North Chungcheong
  - Incheon Clinical Site 102, Incheon
  - Seoul Clinical Site 101, Seoul
  - Seoul Clinical Site 107, Seoul
  - Seoul Clinical Site 108, Seoul
  - Seoul Clinical Site 109, Seoul
  - Seoul Clinical Site 110, Seoul
  - Ulsan Clinical Site 105, Ulsan

IPD SHARING:
Plan to Share IPD: Yes
URL: https://www.ono.co.jp/eng/rd/policy.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 104 subjects determined eligible, 1 had an unknown histological type and excluded.
Groups:
- Squamous Non-small Cell Lung Cancer (NSCLC); Non-squamous Non-small Cell Lung Cancer (NSCLC): In each treatment cycle, patients received an intravenous infusion of nivolumab (ONO-4538) at a dose of 3 mg/kg with 2-week dosing intervals for 6 weeks. Radiological assessments (computed tomography/ magnetic resonance imaging) were conducted every 6 weeks. Patients entered subsequent treatment cycles unless they met discontinuation criteria, including disease progression, unacceptable adverse events, and consent withdrawal. Patients who were discontinued for any of these reasons entered the follow-up phase.
Period: Overall Study
Arm/Group | Squamous Non-small Cell Lung Cancer (NSCLC) | Non-squamous Non-small Cell Lung Cancer (NSCLC)
Started | 45 | 58
Completed | 12 | 15
Not Completed | 33 | 43
Not completed — Did not receive the investigational product | 1 | 2
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Met an exclusion criteria | 0 | 1
Not completed — Adverse Event | 3 | 10
Not completed — Disease progression | 20 | 27
Not completed — Other than above reasons | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Squamous Non-small Cell Lung Cancer (NSCLC); Non-squamous Non-small Cell Lung Cancer (NSCLC): Refer to "Participant Flow".
- Total: Total of all reporting groups
Arm/Group | Squamous Non-small Cell Lung Cancer (NSCLC) | Non-squamous Non-small Cell Lung Cancer (NSCLC) | Total
Number analyzed (Participants) | 44 | 56 | 100
Age, Continuous [Median (Full Range); unit: years] | 69.5 [40 to 80] | 63.5 [29 to 77] | 66.5 [29 to 80]
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 14 | 30 | 44
  65-<75 years | 21 | 20 | 41
  >=75 years | 9 | 6 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 22 | 22
  Male | 44 | 34 | 78
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 44 | 56 | 100
Histology [Count of Participants; unit: Participants]
  Squamous | 44 | 0 | 44
  Adenocarcinoma | 0 | 50 | 50
  Large cell carcinoma | 0 | 1 | 1
  Other | 0 | 5 | 5
Disease stage [Count of Participants; unit: Participants] — Clinical stage was diagnosed according to UICC-TNM classification (7th edition) . Generally, the prognosis becomes worse as the stage progresses.
  Participants
    IIIB | 5 | 1 | 6
    IV | 37 | 54 | 91
    Recurrent | 2 | 1 | 3
Prior treatment for NSCLC: Surgery [Count of Participants; unit: Participants]
  Yes | 9 | 9 | 18
  No | 35 | 47 | 82
Prior treatment for NSCLC: Radiotherapy [Count of Participants; unit: Participants]
  Yes | 11 | 13 | 24
  No | 33 | 43 | 76
Prior treatment for NSCLC-Medication: Platinum-based chemotherapy [Count of Participants; unit: Participants]
  Yes | 44 | 56 | 100
  No | 0 | 0 | 0
Prior treatment for NSCLC-Medication: EGFR-TKI therapy [Count of Participants; unit: Participants] — EGFR-TKI: epidermal growth factor receptor-tyrosine kinase inhibitors.
  Participants
    Yes | 1 | 7 | 8
    No | 43 | 49 | 92
Number of treatment regimens for NSCLC [Count of Participants; unit: Participants]
  1 | 42 | 49 | 91
  2 | 2 | 7 | 9
Smoking history [Count of Participants; unit: Participants]
  Never smoker | 1 | 21 | 22
  Current/former smoker | 43 | 35 | 78
Eastern Cooperative Oncology Group performance status [Count of Participants; unit: Participants] — PS 0 means "fully active, able to carry on all pre-disease performance without restriction" whereas PS 1 means "restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work". Generally, the prognosis worsens as PS worsens.
  Participants
    0 | 6 | 8 | 14
    1 | 38 | 48 | 86
Brain metastasis [Count of Participants; unit: Participants]
  Yes | 10 | 16 | 26
  No | 34 | 40 | 74
EGFR status [Count of Participants; unit: Participants]
  Positive | 1 | 7 | 8
  Negative | 13 | 43 | 56
  Unknown | 30 | 6 | 36

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Centrally Assessed)
Description: Response rate (%) = (Number of subjects whose confirmed best overall response was complete response (CR) or partial response (PR) / Total number of FAS)*100. 95% Confidence interval (CI) was calculated by Wilson method.
Time Frame: Screening phase: Up to 14 days before enrollment.Treatment phase: Day 43 of each cycle or end of treatment phase (up to approximately 10 months).Follow-up phase: 28 days after final dose or for discontinuation occurring 28 or fewer days after final dose.
Population: Full analysis set（FAS): This set was defined as a full group of subjects who were included in safety analysis set, which was defined as group of subjects who were enrolled and received at least one dose of the study drug. This set was used in the primary efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Squamous Non-small Cell Lung Cancer (NSCLC) | Non-squamous Non-small Cell Lung Cancer (NSCLC)
Number analyzed (Participants) | 44 | 56
percentage of participants | 13.6 [6.4 to 26.7] | 19.6 [11.3 to 31.8]

2. Secondary Outcome: Response Rate (Investigator-assessed)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: as for outcome 1
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Squamous Non-small Cell Lung Cancer (NSCLC) | Non-squamous Non-small Cell Lung Cancer (NSCLC)
Number analyzed (Participants) | 44 | 56
percentage of participants | 18.2 [9.5 to 32.0] | 19.6 [11.3 to 31.8]

3. Secondary Outcome: Overall Survival
Description: Overall survival (days) = (the date of death due to any cause) - (the first dose date of investigational product) + 1. 95% CI was calculated by Kaplan-Meier method.
Time Frame: Follow-up phase: Every 6 months after the first day of treatment of the last subject enrolled in the study, until death or study completion.
Population: FAS
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Squamous Non-small Cell Lung Cancer (NSCLC) | Non-squamous Non-small Cell Lung Cancer (NSCLC)
Number analyzed (Participants) | 44 | 56
days | NA [249.0 to NA] — During the period up to the cut-off, 27 (27.0%) out of 100 subjects in the FAS died (fatal) [squamous NSCLC 12 subjects (27.3%), non-squamous NSCLC 15 subjects (26.8%)] and median overall survival could not be estimated. And the upper limit of the 95% CI for the median could not be obtained. There was an insufficient number of participants with events. | NA [291.0 to NA] — During the period up to the cut-off, 27 (27.0%) out of 100 subjects in the FAS died (fatal) [squamous NSCLC 12 subjects (27.3%), non-squamous NSCLC 15 subjects (26.8%)] and median overall survival could not be estimated. And the upper limit of the 95% CI for the median could not be obtained. There was an insufficient number with events.

4. Secondary Outcome: Progression Free Survival (Centrally Assessed)
Description: Progression free survival (days) = (the earlier date of the first documented progressive disease (PD) or death due to any cause) - (the first dose date of investigational product) + 1. 95% CI was calculated by Kaplan-Meier method.
Time Frame: Screening phase: Up to 14 days before enrollment.Treatment phase: Day 43 of each cycle or until central PD was confirmed or data cut-off point.Follow-up phase: Until beginning subsequent treatment for non-small cell lung cancer or PD or recurrence.
Population: FAS
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Squamous Non-small Cell Lung Cancer (NSCLC) | Non-squamous Non-small Cell Lung Cancer (NSCLC)
Number analyzed (Participants) | 44 | 56
days | 67.0 [41.0 to 182.0] | 162.0 [43.0 to 216.0]

5. Secondary Outcome: Duration of Response (Centrally Assessed)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Duration of response (days) = (the date of the first documented PD or death due to any cause after response was confirmed) - (the date of the first confirmed CR or PR) + 1. Median (95% CI) was calculated by Kaplan-Meier method.
Time Frame: Screening phase: Up to 14 days before enrollment.Treatment phase: Day 43 of each cycle or end of treatment phase(up to approximately 10 months).Follow-up phase: Until beginning subsequent treatment for non-small cell lung cancer or PD or recurrence.
Population: FAS
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Squamous Non-small Cell Lung Cancer (NSCLC) | Non-squamous Non-small Cell Lung Cancer (NSCLC)
Number analyzed (Participants) | 44 | 56
days | NA [145.0 to NA] — Median duration of response could not be estimated and the upper limit of the 95% CI for the median could not be obtained. There was an insufficient number of participants with events. | NA [85.0 to NA] — Median duration of response could not be estimated and the upper limit of the 95% CI for the median could not be obtained. There was an insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: From the start of the first dose of the investigational product to 28 days after the final dose or discontinuation, occurring 28 or fewer days after the final dose, or data cut-off point (June 2, 2015), whichever occurs first. Adverse events will be monitored and assessed before each dose and as needed based on clinical symptoms. Total assessment period: up to 10 months per participant.
Description: The analysis was performed on SAS, which was defined as group of subjects who received at least one dose of the study drug. Adverse Events (AEs) were analyzed based on treatment emergent AEs (TEAEs), defined as any event not present prior to initiation of study drug that first appeared following exposure to study drug or any event already presented that worsened relative to the pre-treatment state following the treatment. All-Cause Mortality was defined as incidence of TEAEs leading to death.
Arm/Group | Squamous Non-small Cell Lung Cancer (NSCLC) | Non-squamous Non-small Cell Lung Cancer (NSCLC)
All-Cause Mortality (participants affected / at risk) | 12/44 | 15/56
Serious Adverse Events (participants affected / at risk) | 20/44 | 17/56
Other Adverse Events (participants affected / at risk) | 24/44 | 36/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Squamous Non-small Cell Lung Cancer (NSCLC) (N=44) | Non-squamous Non-small Cell Lung Cancer (NSCLC) (N=56)
Angina unstable (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Pneumonia (Infections and infestations) | 5 | 4
Sialoadenitis (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infarction (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Squamous Non-small Cell Lung Cancer (NSCLC) (N=44) | Non-squamous Non-small Cell Lung Cancer (NSCLC) (N=56)
Constipation (Gastrointestinal disorders) | 8 | 11
Diarrhoea (Gastrointestinal disorders) | 6 | 2
Dyspepsia (Gastrointestinal disorders) | 5 | 5
Nausea (Gastrointestinal disorders) | 6 | 6
Asthenia (General disorders) | 3 | 4
Chest discomfort (General disorders) | 1 | 3
Chest pain (General disorders) | 6 | 5
Chills (General disorders) | 2 | 4
Fatigue (General disorders) | 7 | 11
Influenza like illness (General disorders) | 2 | 3
Pain (General disorders) | 4 | 3
Pyrexia (General disorders) | 7 | 8
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 18 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 6
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 5
Dizziness (Nervous system disorders) | 4 | 6
Headache (Nervous system disorders) | 2 | 6
Anxiety (Psychiatric disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 4 | 5
Dysuria (Renal and urinary disorders) | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 15
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 12
Rash (Skin and subcutaneous tissue disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this tiral prior to submission for publication/presentation.

DOCUMENTS (2):
  • Study Protocol (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/17/NCT02175017/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT02175017/SAP_001.pdf